CLINICAL TRIAL: NCT03542162
Title: Patching Retinal Breaks With Healaflow in 27G Vitrectomy for the Treatment of Rhegmatogenous Retinal Detachment
Brief Title: Healaflow Patch for the Treatment of Rhegmatogenous Retinal Detachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Zhenchuan Zheng, Principal investigator, Tianjin Medical University Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-KY18
Record Dates: First submitted 2018-05-17; First posted 2018-05-31 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: Healaflow; Rhegmatogenous retinal detachment; 27-gauge Pars plana vitrectomy; Minimally invasive surgery; Complications

STUDY DESIGN:
Intervention Model Description: All patients who meet the criteria and agree to paticipate in the clinical study, will be enrolled to this study after signing informed consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healaflow group (Experimental): The Healaflow group consists of patients with primary RRD, but exclude proliferative vitreoretinopathy grade C or more, dialysis, retinoschisis, eyes with secondary RRD, significant corneal or lens opacity precluding vitrectomy, giant retinal tears, a follow-up period of less than 3 months, and visual loss from causes other than RRD.
  Interventions: Biological: Healaflow

INTERVENTIONS:
Biological: Healaflow — For the RRD patients, after 27G PPV, air-liquid exchange and endolaser photocoagulation around the tear(s), Healaflow is going to be fully covered on the surface of all retinal tears using 27G needle, the amount of Healaflow injection was determined according to the size of tears.

SUMMARY:
To report the surgical results of primary rhegmatogenous retinal detachment (RRD) repaired by 27G pars plana vitrectomy (PPV) combined with Healaflow patch and air tamponade, and do not need prone position postoperation.

DETAILED DESCRIPTION:
To improve the success rates of pars plana vitrectomy(PPV) which is the most common surgical procedure for the repair of primary rhegmatogenous retinal detachment (RRD) and to avoid silicon oil tamponade and face-down position, all eyes enrolled into this clinical trail undergo 27G PPV combined with Healaflow patch and air tamponade which do not need face-down position in the postoperative period. Healaflow® (Anteis S.A., Plan Les Ouates, Switzerland) consists of over 97% water, sodium hyaluronic acid (22.5 mg/ml) of nonanimal origin cross-linked with BDDE (1.4-Butanediol diglycidyl ether), and phosphate- and NaCl-salts to maintain a physiological pH (7.0) and osmolarity (305 mOsm/kg).

At the time of study enrollment, physical examinations, best-corrected visual acuity (BCVA), intraocular pressure(IOP) will be measured and fundoscopy, OCT, B-ultrasound will be performed.

The patients are going to be followed up for at least 3 months, the main outcome measures are postoperative primary and final anatomic outcome, BCVA and complications.

ELIGIBILITY:
Inclusion Criteria: - patients with primary RRD

Exclusion Criteria: - proliferative vitreoretinopathy grade C or more, dialysis, retinoschisis, eyes with secondary RRD, significant corneal or lens opacity precluding vitrectomy, giant retinal tears, a follow-up period of less than 3 months, and visual loss from causes other than RRD

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
postoperative anatomic outcome | baseline to 3 months post-surgery
  fundus retina examination through ophthalmoscope, fundus image, B ultrosound

SECONDARY OUTCOMES:
BCVA | baseline to 3 months post-surgery
  BCVA using a Landolt C acuity chart method
postoperative complications | baseline to 3 months post-surgery
  postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Li, MD, PhD, Principal Investigator — Tianjin Medical University Eye Hospital

IPD SHARING:
Plan to Share IPD: No